CLINICAL TRIAL: NCT00061867
Title: A Dose Escalation, Pharmacokinetics, and Safety Study of Doxorubicin Encapsulated in Temperature Sensitive Liposomes Released Through Microwave Therapy in the Treatment of Prostate Cancer
Brief Title: Liposomal Doxorubicin and Thermal Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imunon (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CELSION-10302101; CDR0000301761 (Registry Identifier: PDQ (Physician Data Query)); RPCI-DS-0228
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2005-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diathermy

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin hydrochloride
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, use different ways to stop tumor cells from dividing so they stop growing or die. Microwave thermotherapy kills tumor cells by heating them to several degrees above body temperature. Combining liposomal doxorubicin with microwave thermotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of liposomal doxorubicin when given together with microwave thermotherapy in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of doxorubicin HCl liposome released through thermal microwave therapy in patients with adenocarcinoma of the prostate.
* Determine the pharmacokinetics and biodistribution profile of this drug in these patients.
* Determine the safety profile and dose-limiting toxicity of this drug in these patients.
* Determine the clinical response in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive doxorubicin HCl liposome IV over 30 minutes. Patients then undergo a 60-minute course of prostate thermotherapy. Treatment may repeat every 28-42 days for up to 6 courses, at the discretion of the physician.

Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 8, 15, 30, and 90 days.

PROJECTED ACCRUAL: Approximately 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Rising prostate-specific antigen AND radiographic evidence of extraprostatic prostate cancer by bone scan, CT scan, prostascint scan, or MRI

PATIENT CHARACTERISTICS:

Age

* 40 and over

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic

* Bilirubin normal
* AST normal
* Alkaline phosphatase normal
* No acute or chronic liver disease

Renal

* Creatinine less than 1.5 times upper limit of normal

Cardiovascular

* Ejection fraction at least 50% by MUGA
* EKG normal
* No myocardial infarction or cerebral vascular accident within the past 6 months
* No life threatening cardiac arrhythmias
* No congestive heart failure
* No cardiac pacemaker
* No peripheral arterial disease with intermittent claudication or Leriches syndrome (i.e., claudication of the buttocks or perineum)

Other

* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No sperm donation during and for 3 months after study participation
* Not febrile
* No interest in future fertility or fathering children
* No significantly decreased pain response
* No severe urethral stricture
* No protruding median lobe resulting in a "ball-valve" type of obstruction at the bladder neck
* No major psychiatric illness that would prevent informed consent
* No major psychiatric illness that required inpatient treatment within the past 3 months
* No psychological, family, sociological, or geographic condition that would preclude study compliance
* No allergy to eggs or egg products
* No urinary or prostatic infection
* No full urinary retention
* No penile or urinary sphincter implant
* No metallic implants in the pelvic or femoral area
* No other serious medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent live vaccines

Chemotherapy

* No prior anthracycline
* No concurrent streptozocin

Endocrine therapy

* No concurrent hormonal therapy (except luteinizing hormone-releasing hormone analog)
* No concurrent glucocorticoids administered at more than physiologic replacement doses (other than as an antiemetic)

Radiotherapy

* Not specified

Surgery

* More than 3 months since prior major surgery

Other

* No prior therapy that resulted in permanent reduction of pain response (e.g., prior surgery, regional or local anesthetic)
* No concurrent PC-SPES
* No concurrent cyclosporine, phenobarbital, or phenytoin

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Doren, RN, Study Chair — Imunon
Locations (2):
- United States (2):
  - Regional Urology, L.L.C., Shreveport, Louisiana
  - Grand Strand Urology LLP, Myrtle Beach, South Carolina